CLINICAL TRIAL: NCT02525640
Title: Hearing Handicap in Patients With Single Sided Deafness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants recrui
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Rachel Knappett, Specialist Audiologist, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 108402; A092833 (Other: Addenbrookes Hospital, Cambridge)
Record Dates: First submitted 2014-09-03; First posted 2015-08-17 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Hearing Loss
Keywords: Single sided hearing loss; Single sided deafness; Hearing loss music appreciation
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hearing Aid (Experimental): CROS hearing aid
  Interventions: Device: Hearing Aid

INTERVENTIONS:
Device: Hearing Aid — Hearing aid comparison
  Other Names: Phonak Nathos S+ Micro Wireless CROS aid; Oticon Spirit Zest Wired CROS aid

SUMMARY:
Single sided deafness (SSD) refers to asymmetrical hearing loss, where there is a significant worsening of hearing in one ear compared to the other.

In Cambridge, the investigators see large numbers of patients with SSD caused by vestibular schwannomas, due to their affiliation with the Neuro-Otology Department, with over 100 new SSD patients being referred every year.

Only a small number of studies have explored hearing handicap for those with SSD, and music appreciation has not been investigated, to the best of the investigators knowledge, in this patient group.

In the limited number of studies conducted on those with single sided deafness, often only one or two outcome measures have been used, or the patient group has been small. The investigators have a large group of patients with a wide range of aetiologies who have completed several questionnaires as part of their treatment in the single sided deafness clinic and the investigators would like to analyse these data.

At present there are different devices available on the NHS for the management of SSD and many studies have explored benefits of Bone Anchored Hearing Aids (BAHA). There is an under-representation of studies looking specifically at CROS aid devices which is relevant given the cost differences involved between devices.

Study goals and objectives

* To find out what factors drive hearing handicap in SSD patients by analysing the results of several different well validated hearing handicap questionnaires
* To find out whether or not it is possible to change hearing handicap in this patient group by looking to see if there is an improvement in questionnaire scores post treatment.
* The investigators will also look at a sub-group who will be fitted with both traditional wired CROS aids and more up-to-date wireless aids which have been funded through a research grant, in order to assess whether these are more beneficial.
* The investigators will use a new questionnaire developed in-house to further explore the impact of single sided deafness on music appreciation.

DETAILED DESCRIPTION:
SSD can lead to:

* Reduction in spatial hearing
* Significant difficulty in background noise and social situations
* Exhaustion from the extra effort required to hear
* Reduced confidence
* Reduced ability to enjoy music
* Isolation
* An emotional burden linked to the onset of the hearing loss and associated symptoms

The investigators have established a specialised clinic to address the consequences of SSD, and assess treatment options including the provision of counselling and wired CROS (Contralateral Routing of Signal) hearing aids.

The investigators use a range of questionnaires, completed pre and post treatment, to assess outcomes and would like to analyse this data to see what drives handicap and whether there is any observable improvement post treatment. The investigators would like to find out more about the impact of SSD on patients' ability to enjoy music and propose to do this using a questionnaire developed in-house.

The investigators have been awarded a grant to fit some of their patients with wireless CROS aids, which are not routinely available under the NHS in Cambridge, but are widely available in other areas and in the commercial sector.

The investigators will utilise retrospective data in the form of questionnaires completed by SSD patients attending the Audiology clinic between 2009 and 2012. Prospective data will also be collected and from existing SSD patients, to whom the investigators intend to post the music appreciation questionnaire, or ask them to complete in clinic.

A prospective cross over design study will compare wired and wireless CROS hearing aids in 13 new patients a cross-over design trial to investigate whether residual handicap and satisfaction are any better with these devices than with standard wired versions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who attend the single sided deafness clinic.
* Must have either no recordable hearing threshold levels on one side or a significant asymmetry.
* The 13 CROS aid trial patients must be post-operative vestibular schwannoma patients with an audiological 'dead ear' on the affected side.

Exclusion Criteria:

* Patients unable to give informed consent
* Patients under 18 years of age
* For the CROS aid trial, patients with any aetiology other than vestibular schwanomma, pre-operative vestibular schwanomma patients or vestibular schwanomma patents who still have residual hearing in the affected ear.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08-01 (Estimated); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Abbreviated hearing aid benefit profile (APHAB) | 180 days
  Hearing aid benefit questionnaire
Speech and spatial qualities of hearing (SSQ) | 180 days
  Hearing aid benefit questionnaire
Tinnitus handicap inventory (THI) | 180 days
  Tinnitus questionnaire
Hearing handicap inventory (HHI) | 180 days
  Hearing aid benefit questionnaire
Hospital anxiety and depression scale (HADS) | 180 days
  Anxiety and depression questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Smith, MSc, Principal Investigator — Addenbrooke's Hospital, Cambridge, UK
Locations (1):
- Cambridge University Hospital NHS Trust, Audiology department, Cambridge, Cambridgeshire, United Kingdom